CLINICAL TRIAL: NCT00960401
Title: Pilot Study "A Study of Atherosclerosis in Patients After Radiation Treatment for Breast Cancer"
Brief Title: A Study of Atherosclerosis in Patients After Radiation Treatment for Breast Cancer
Acronym: ABCART
Status: Completed | Type: Observational
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 05018
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Results first posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-02

CONDITIONS: Atherosclerosis
Keywords: coronary calcium scoring; breast cancer patients; radiation treatment
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- cardiac counseling: 10 left sided breast cancer patients 10 right sided breast cancer patients
- coronary artery evaluation: 10 left sided breast cancer 10 right sided breast cancer

SUMMARY:
The purpose of this study is to compare plaque burden in the coronary and carotid arteries 5 years after adjuvant radiotherapy in women with right sided breast cancer vs left sided breast cancer.

DETAILED DESCRIPTION:
This study reviews case series of patients with a history of breast cancer treated with radiotherapy for at least five years. The study measures atherosclerosis by using coronary and carotid artery calcium scoring.

ELIGIBILITY:
Inclusion Criteria:

* women dx with ductal carcinoma in situ or breast cancer, stage 0 to stage IIIc, who received conservative surgery and radiotherapy at least 5 years ago
* less than or equal to age 60

Exclusion Criteria:

* hx of coronary disease prior to tx of ductal carcinoma in situ or breast cancer

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: breast cancer patients after radiation treatment
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-08; Primary Completion 2007-05 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hindenburg, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

REFERENCES:
- [Background] Chang M, Suh J, Kirtani V, Dobrescu A, Haas J, Zeldis S, Shayani S, Hindenburg AA. Coronary Calcium Scanning in Patients after Adjuvant Radiation for Early Breast Cancer and Ductal Carcinoma In situ. Front Oncol. 2013 Sep 25;3:253. doi: 10.3389/fonc.2013.00253. eCollection 2013. PMID 24093087

RESULTS

PARTICIPANT FLOW:
Groups:
- Coronary Artery Evaluation Left Side Breast Cancer: 9 left sided breast cancer
- Coronary Artery Evaluation Right Side Breast Cancer: 11 right sided breast cancer
Period: Overall Study
Arm/Group | Coronary Artery Evaluation Left Side Breast Cancer | Coronary Artery Evaluation Right Side Breast Cancer
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Age 60 years or younger at time of radiatiion to chest wall. All subjects had radiation at least 5 years prior to enrollment. Patients with clinical symtoms of CAD were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Coronary Artery Evaluation Left Side Breast Cancer | Coronary Artery Evaluation Right Side Breast Cancer | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Analyzed for Coronary Calcium Burden by AGS
Description: Number of participants who received a coronary calcium scan.
Time Frame: Year 5 Post-Initiation of Radiotherapy
Measure: Count of Participants; unit: Participants
Groups:
- Coronary Artery Evaluation Right Side Breast Cancer: 11 right side breast cancer
Arm/Group | Coronary Artery Evaluation Left Side Breast Cancer | Coronary Artery Evaluation Right Side Breast Cancer
Number analyzed (Participants) | 9 | 11
Participants | 9 | 11

ADVERSE EVENTS:
Groups:
- Coronary Artery Evaluation: 9 left sided breast cancer 11right sided breast cancer
Arm/Group | Coronary Artery Evaluation
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes